CLINICAL TRIAL: NCT00707200
Title: Clinical Outcomes in Pediatric Plasmodium Falciparum Malaria According to Host Cytoadherence Factors
Brief Title: The Cytoadherence in Pediatric Malaria (CPM) Study
Acronym: CPM
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Christine Cserti-Gazdewich, University Health Network
Other Study IDs: 07-0548-AE; HS 356; ISBT 777531237
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2009-07

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: severe malarial anemia (SMA); cerebral malarial (CM); lactic acidosis; hyperparasitemia; respiratory distress; hypoxia; death; transfusion
MeSH Terms: conditions — Malaria, Falciparum; Acidosis, Lactic; Dyspnea; Hypoxia; Death

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Freshly frozen citrated plasma aliquots, frozen spun red cell pellets, and whole blood blots onto nucleic acid storage cards (Whatman FTA).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Cases: Severe inpatient malaria, survivors or decedents. Severe malaria consists of any one or combination of severe malarial anemia (SMA), cerebral malaria (CM), lactic acidosis (LA), or a respiratory distress syndrome with hypoxia.
- 2: Controls: Controls consist of mildly-affected children with P falciparum malaria who are either managed as inpatients or outpatients.

SUMMARY:
The purpose of this study is to determine the importance of key blood group molecules in the clinical outcome of Plasmodium falciparum malaria infection in children.

DETAILED DESCRIPTION:
Every year, nearly 2 million children die from infection with Plasmodium falciparum malaria. When red blood cells (RBC) become infected with malaria, a sticky parasite-derived knob protein, termed PfEMP-1, erupts on the RBC surfaces. PfEMP-1 attaches to several blood group molecules, including those found on other RBC, on blood vessels, and on the cells that normally help to stop bleeding (platelets). The cellular sticking results in a dangerous interruption in blood flow to vital organs, causing brain injury (cerebral malaria), systemic shock (lactic acidosis), and death. Depending on an individual's inherited blood groups of relevance, adhesion may be extensive or limited. In the laboratory, PfEMP-1 adheres to RBCs via the A or B (but not the O) antigens of the ABO blood group system, and to platelets and blood vessels via platelet glycoprotein IV (CD36) and ICAM-1. Consistent with the expected evolutionary advantage of being deficient in these binding targets, blood type O and low-expression of CD36 are found more frequently among Africans. The "Cytoadherence in Pediatric Malaria" (CPM) project is determining the distribution of adhesive blood group molecules in a cohort of 2000 Ugandan children according to the extent of malaria severity and death, and thus their ultimate clinical and evolutionary significance in malarial survival. This knowledge may serve as the grounds for developing targeted cytoadhesion-interruption therapies in our fight against malaria.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Plasmodium falciparum malaria infection

Exclusion Criteria:

* HIV or significant malnutrition

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children, age 6 months to 12 years, with symptomatic malaria and (asexual) Plasmodium falciparum parasitemia.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Combined severe morbidity & mortality | Discharge

SECONDARY OUTCOMES:
Laboratory indices of potential cytoadhesion (lactate, cell counts) | Presentation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolette Nabukeera-Barungi, MBChB, MMEd, Study Director — Mulago Hospital/Makerere University (lead local investigator)
Locations (1):
- Mulago Hospital Acute Care Unit & Makerere University Department of Paediatrics & Child Health, Kampala, Uganda

REFERENCES:
- [Background] Cserti CM, Dzik WH. The ABO blood group system and Plasmodium falciparum malaria. Blood. 2007 Oct 1;110(7):2250-8. doi: 10.1182/blood-2007-03-077602. Epub 2007 May 14. PMID 17502454
- [Result] Cserti-Gazdewich CM, Dzik WH, Dorn ME, Quagliaroli RO, Xu S, Ssewanyana I, Nayyar R, Preffer FI. Quantitation of CD36 (platelet glycoprotein IV) expression on platelets and monocytes by flow cytometry: application to the study of Plasmodium falciparum malaria. Cytometry B Clin Cytom. 2009 Mar;76(2):127-34. doi: 10.1002/cyto.b.20443. PMID 18671254
- [Derived] Cserti-Gazdewich CM, Dhabangi A, Musoke C, Ssewanyana I, Ddungu H, Nakiboneka-Ssenabulya D, Nabukeera-Barungi N, Mpimbaza A, Dzik WH. Inter-relationships of cardinal features and outcomes of symptomatic pediatric Plasmodium falciparum MALARIA in 1,933 children in Kampala, Uganda. Am J Trop Med Hyg. 2013 Apr;88(4):747-756. doi: 10.4269/ajtmh.12-0668. Epub 2013 Jan 28. PMID 23358640